CLINICAL TRIAL: NCT00935155
Title: Effectiveness of Acupuncture as an Adjunct to Rehabilitation After Knee Arthroplasty. A Randomized Controlled Trial.
Brief Title: Effectiveness of Acupuncture as an Adjunct to Rehabilitation After Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Back and Rehabilitation Center, Copenhagen (Other Government)
Responsible Party: Principal Investigator, Tom Petersen, Physical Therapist, Back and Rehabilitation Center, Copenhagen
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: VIFAB-727-44-2007
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Total Knee Replacement
Keywords: exercise therapy; Knee arthroplasty; Acupuncture Analgesia; Arthroplasty, Replacement, Knee; rehabilitation
MeSH Terms: interventions — Acupuncture Therapy; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): Acupuncture in combination with exercise therapy
  Interventions: Procedure: Acupuncture
- exercises (Active Comparator): Coordination, mobilizing, endurance, strength
  Interventions: Procedure: exercises

INTERVENTIONS:
Procedure: Acupuncture — Westerns style acupuncture. Twice a week for 12 weeks
  Arms: Acupuncture
Procedure: exercises — Coordination, mobilizing, endurance, strength
  Arms: exercises

SUMMARY:
No randomized trials have tested the effectiveness of acupuncture as a supplement to rehabilitation after total knee replacement. Studies from related fields, however, have shown reduction of symptoms as a result of acupuncture treatment in patients with knee pain caused by severe osteoarthritis in the knee. Furthermore, studies have reported that the need of pain medication was lower when acupuncture treatment was performed immediately after knee surgery.

The aim of this study is to test whether acupuncture can reduce pain and improve disability as a supplement to rehabilitation after total knee replacement.

One hundred and seventy patients will be allocated by drawing lots to either a treatment group receiving exercise therapy and acupuncture or a group receiving exercise therapy alone. Treatment will start 3 weeks after surgery at the latest.

Outcome of treatments will be measured at completion of treatment and at 3 months follow-up by pain- and disability questionnaires as well as the recording of walking capacity.

ELIGIBILITY:
Inclusion Criteria:

* Hemi- or total knee arthroplasty.
* 18 - 70 years of age.

Exclusion Criteria:

* Concurrent diseases that compromises treatment, i.e.hip disease, rheumatoid arthritis, migraine).
* Bleeding disorders.
* Heart disease or use of pacemaker.
* Lack of patient cooperation, i.e. psychological disorders, alcoholism, problems with language).
* Infection.

Exclusion criteria during intervention:

* Infection.
* Cicatrice-burst.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
pain | 3 months after treatment

SECONDARY OUTCOMES:
disability | 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tom Petersen, PT, PhD, Principal Investigator — Back and Rehabilitation Center, Copenhagen
Locations (1):
- Back and Rehabilitation Center Copenhagen, Copenhagen, Copenhagen, Denmark